CLINICAL TRIAL: NCT00917761
Title: Entecavir and Peginterferon Alfa-2a Sequential Therapy Versus Peginterferon Alfa-2a Monotherapy for HBeAg Negative Chronic Hepatitis B
Brief Title: Entecavir and Pegasys Sequential Therapy Versus Pegasys for HBeAg Negative Chronic Hepatitis B
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 950924
Record Dates: First submitted 2009-06-08; First posted 2009-06-10 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2012-12

CONDITIONS: Hepatitis B, Chronic
Keywords: Hepatitis B, chronic; Peginterferon alfa-2a; Entecavir
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir; peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Entecavir and peginterferon (52 weeks) (Experimental): Entecavir 0.5 mg/day po at week 1-4 Peginterferon alfa-2a 180 ug/week sc at week 5-52
  Interventions: Drug: Entecavir and peginterferon (Pegasys) (52 weeks)
- Peginterferon (96 weeks) (Experimental): Peginterferon alfa-2a 180 ug/week sc at week 1-96
  Interventions: Drug: Peginterferon (Pegasys) (96 weeks)
- Peginterferon (48 weeks) (Active Comparator): Peginterferon alfa-2a 180 ug/week sc at week 1-48
  Interventions: Drug: Peginterferon (Pegasys) (48 weeks)

INTERVENTIONS:
Drug: Entecavir and peginterferon (Pegasys) (52 weeks) — Entecavir 0.5 mg/day po at week 1-4 Peginterferon alfa-2a 180 ug/week sc at week 5-52
  Other Names: Entecavir (Baraclude)0.5 mg/day po at week 1-4; Peginterferon alfa-2a (Pegasys) 180 ug/week sc at week 5-52
  Arms: Entecavir and peginterferon (52 weeks)
Drug: Peginterferon (Pegasys) (96 weeks) — Peginterferon alfa-2a 180 ug/week sc at week 1-96
  Other Names: Peginterferon alfa-2a (Pegasys) 180 ug/week sc at week 1-96
  Arms: Peginterferon (96 weeks)
Drug: Peginterferon (Pegasys) (48 weeks) — Peginterferon alfa-2a 180 ug/week sc at week 1-48
  Other Names: Peginterferon alfa-2a (Pegasys) 180 ug/week sc at week 1-48
  Arms: Peginterferon (48 weeks)

SUMMARY:
Currently, peginterferon alfa-2a or oral nucleos(t)ides are approved for the treatment with HBeAg negative CHB, with the overall ALT normalization and HBV viral suppression far from satisfactory. Therefore, efforts on the various combinations with the currently available drugs are needed to improve the overall response rates. The simultaneous combination therapy with oral nucleoside and peginterferon alfa-2a from large-scaled randomized trials did not show a superior response rate over peginterferon alfa-2a monotherapy. Recently, sequential monotherapy with lamivudine for the first 4 weeks, followed by weekly peginterferon alfa-2a has shown favorable HBeAg seroconversion rate over peginterferon alfa-2a monotherapy, based on the assumption that early viral suppression by lamivudine can restore the immune function to facilitate the later immunomodulatory response by peginterferon alfa-2a. Furthermore, prior studies using 24 months of standard interferon alfa showed better ALT normalization and HBV suppression rates to 12 months of therapy. With the recent introduction of entecavir, the more potent oral nucleoside with few drug resistance, sequential monotherapy with entecavir can potently suppress HBV DNA with 4 weeks of treatment, which may facilitate the response of peginterferon alfa-2a to achieve HBV viral suppression. Therefore, we aimed to conduct a placebo controlled randomized control trial to evaluate if adding entecavir early in the course of therapy or extending the treatment duration of peginterferon alfa-2a can improve the treatment response.

DETAILED DESCRIPTION:
Chronic hepatitis B (CHB) is prevalent in the world, with estimated chronic carriers of 350 millions worldwide. Currently, peginterferon alfa-2a or oral nucleos(t)ides are approved for the treatment with HBeAg negative CHB, with the overall ALT normalization and HBV viral suppression far from satisfactory. Therefore, efforts on the various combinations with the currently available drugs are needed to improve the overall response rates. The simultaneous combination therapy with oral nucleoside and peginterferon alfa-2a from large-scaled randomized trials did not show a superior response rate over peginterferon alfa-2a monotherapy. Recently, sequential monotherapy with lamivudine for the first 4 weeks, followed by weekly peginterferon alfa-2a has shown favorable HBeAg seroconversion rate over peginterferon alfa-2a monotherapy, based on the assumption that early viral suppression by lamivudine can restore the immune function to facilitate the later immunomodulatory response by peginterferon alfa-2a. Furthermore, prior studies using 24 months of standard interferon alfa showed better ALT normalization and HBV suppression rates to 12 months of therapy. With the recent introduction of entecavir, the more potent oral nucleoside with few drug resistance, sequential monotherapy with entecavir can potently suppress HBV DNA with 4 weeks of treatment, which may facilitate the response of peginterferon alfa-2a to achieve HBV viral suppression. Therefore, we aimed to conduct a placebo controlled randomized control trial to evaluate if adding entecavir early in the course of therapy or extending the treatment duration of peginterferon alfa-2a can improve the treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis B (presence of HBsAg > 6 months) with anti-HBe persistence and abscence of HBeAg for more than 3 months
* Age older than 18 years
* HBV DNA > 2,000 IU/mL for more than 2 occasions
* Serum ALT levels between 2 to 10 folds the upper limit of normal (ULN)
* A liver biopsy compatible with chronic hepatitis B

Exclusion Criteria:

* Anemia (hemoglobin < 13 gram per deciliter for men and < 12 gram per deciliter for women)
* Neutropenia (neutrophil count <1,500 per cubic milliliter)
* Thrombocytopenia (platelet <90,000 per cubic milliliter)
* Co-infection with hepatitis B virus (HBV), hepatitis D virus (HDV) or human immunodeficiency virus (HIV)
* Chronic alcohol abuse (daily consumption > 20 gram per day)
* Decompensated liver disease (Child-Pugh class B or C)
* Serum creatinine level more than 1.5 times the upper limit of normal
* Autoimmune liver disease
* Neoplastic disease
* An organ transplant
* Immunosuppressive therapy
* Poorly controlled autoimmune diseases, pulmonary diseases, cardiac diseases, psychiatric diseases, neurological diseases, diabetes mellitus
* Evidence of drug abuse
* Unwilling to have contraception
* Known allergic reaction to entecavir or peginterferon alfa-2a
* Unwilling to sign inform consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2007-02; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
HBV virologic response (HBV DNA < 2,000 IU/mL) 6 months after the cessation of treatment | 2.5 years

SECONDARY OUTCOMES:
ALT normalization rate (ALT < 40 IU/L) 6 months after the cessation of treatment | 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Chen-Hua Liu, MD, Study Chair — National Taiwan University Hospital; Jia-Horng Kao, MD, PhD, Principal Investigator — National Taiwan University Hospital; Shih-Jer Hsu, MD, Principal Investigator — National Taiwan University Hosptial, Yun-Lin Branch; Chih-Lin Lin, MD, Principal Investigator — Ren-Ai Branch, Taipei City Hospital; Cheng-Chao Liang, MD, Principal Investigator — Far Eastern Memorial Hospital; Ching-Sheng Hsu, MD, Principal Investigator — Buddhist Tzu Chi General Hospital; Sheng-Shun Yang, MD, PhD, Principal Investigator — Taichung Veterans General Hospital
Locations (6):
- Taiwan (6):
  - National Taiwan University Hosptial, Yun-Lin Branch, Douliu
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Buddhist Tzu Chi General Hospital, Taipei
  - Far Eastern Memorial Hospital, Taipei
  - Ren-Ai Branch, Taipei Municipal Hospital, Taipei